CLINICAL TRIAL: NCT02377791
Title: Impact of CYP3A5 Genetic Polymorphisms on Tacrolimus Concentration and Transplant Outcomes During The Early Stage Post-Transplantation in Thai Kidney Transplant Recipients
Brief Title: Impact of CYP3A5 Gene Polymorphisms on Tacrolimus Concentrations and Outcomes in Thai Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Rama 07-57-16
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Kidney Transplant
Keywords: tacrolimus; Cytochrome P-450 CYP3A; Kidney transplant; FK506; Prograf; Rejection; Gene Polymorphism
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA for polymorphism CYP3A5
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: SNP: CYP3A5 gene polymorphisms — Evaluate impact of CYP3A5*1/*1 vs CYP3A5*1/*3 or CYP3A5*3/*3

SUMMARY:
Tacrolimus is a drug used commonly in kidney transplant patients to prevent graft rejection. Tacrolimus acts in a very narrow range in the blood for its optimum activity. If the levels are too high, there is a risk of kidney injury, whereas, if the levels are too low there is a higher risk of rejection and graft loss. Genetic differences in the gene coding for the enzyme cytochrome P450 (CYP3A5), which is responsible for breaking down active tacrolimus can contribute to variations in blood levels of tacrolimus among different individuals taking the same dose of the drug. Certain genetic types lead to low concentrations, whereas certain genetic types can lead to high levels. The proportion of individuals with different types of genetic variations differ among different ethnic populations. Limited data are available in Thai subjects or on the risk have having certain types of genetic variations on the risk of rejection.

This study aims to compare the effects of different types of CYP3A5 gene variations on Tacrolimus drug levels and risk of acute rejection in Thais.

DETAILED DESCRIPTION:
Rationale important theory or hypothesis:

Tacrolimus, a potent calcineurin inhibitor, is commonly used in kidney transplant patients worldwide. Tacrolimus has a narrow therapeutic index. Overdosing increases the risk of dose-related adverse drug reactions and infections, whereas underdosing increases the risk of rejection and graft loss. In addition, achieving therapeutic tacrolimus levels is complicated by high intra- and inter-individual pharmacokinetic variability of the drug. Though, the source of pharmacokinetic variability of tacrolimus is not fully understood. It is known that the inter-individual variation in metabolism of tacrolimus is at least partly due to differences in expression of the cytochrome P450 (CYP) 3A5 enzyme, one of the key proteins involved in tacrolimus systematic clearance.

Mutations due to single nucleotide polymorphism (SNP) of the gene encoding CYP 3A5 have been demonstrated to affect their expression. Among CYP3A5 alleles, CYP3A5*1 has been found to be the main allele associated with CYP 3A5 expression, whereas the mutant allele CYP3A5*3 prevents expression of the enzyme. Several studies have shown that this mutation affects the dosing of tacrolimus.

The frequency of CYP3A5 SNP varies among different ethnic populations . In a small study in Thais, the frequency of , CYP3A5*1/*1 genotyping was identified in 20.6% of patients, CYP3A5*1/*3 in 35.3% and CYP3A5*3/*3 in 44.1%.

To the best of our knowledge, there is no previous study on the impacts of the CYP 3A5 genetic polymorphisms on tacrolimus blood concentration and acute rejection rate during the very early stage post-transplantation in Thai kidney transplant recipients. Evaluation of CYP3A5 polymorphisms may be helpful in determining an appropriate starting dose, timely achieving target levels, and improving outcomes of tacrolimus-based therapy in this group of patients.

Therefore, we are to determine the impacts of CYP 3A5 genetic polymorphisms on tacrolimus trough blood concentration during the first post-operative week and acute rejection rate at 3-month post-transplantation comparing between CYP3A5 expressers (CYP3A5*1 homozygotes or heterozygotes) and CYP3A5 non-expressers (CYP3A5*3 homozygotes).

Methods:

Study population:

This retrospective analytical study will be performed at Ramathibodi hospital, Bangkok, Thailand. Thai recipients who underwent kidney transplantation between January 2011 and December 2013.

Data collection:

Demographics and clinical data will be gathered from the medical files and records. Blood samples will be collected for determination of genotypes of CYP3A5, other metabolic enzymes and transport proteins with respect to their corresponding effects on the pharmacokinetics of tacrolimus.

Approval for this study will be obtained from the ethics committee of Ramathibodi hospital, Faculty of Medicine, Mahidol University.

Number of samples:

According to the study of Sang-Il Min, et al , the effect of CYP3A5*1 allele with early acute rejection and graft function in patients with kidney transplants who received tacrolimus. CYP3A5 expressers (n=29) had the mean trough concentration to dose ratio of 127.09 ± 69.40 ng/mL/mg/kg. While CYP3A5 non-expressers (n=33) had the mean trough concentration to dose ratio of 220.99 ± 108.95 ng/mL/mg/kg on day 10 after kidney transplantation.

The sample size is estimated using the formula: n/group=2(Zα + Zβ)2σ2/(µ1-µ2)2 Given dose adjusted Co of Tac among expressor µ1= 127.09±69.40 and the different at least 25% would have clinical significant so the absolute different was 30. Calculated sample size was at least 85 patients per group so the total subjects would be at least 170 patients.

Ref. Transplantation 2010;90: 1394-1400

Statistical analysis:

Differences in genotype will be assessed using SPSS version 17.0 software for chi square or Mann-Whitney U tests.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplantation between January 2011 and December 2013
2. Received two divided daily doses of tacrolimus in their initial regimen for prevention of allograft rejection
3. Informed consent

Exclusion Criteria:

1. multiple organ transplantation
2. hyperacute rejection
3. non-functioning graft,
4. ABO incompatible kidney transplantation
5. severe liver function or hypoalbuminemia (serum albumin <3 g/dl)
6. severe gastrointestinal disorders that could interfere with their ability to absorb oral medications
7. patients whose recorded data is incomplete;
8. Receiving other medications that can significantly interfere with tacrolimus pharmacokinetics (except methylprednisolone and prednisolone)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai recipients who underwent kidney transplantation between January 2011 and December 2013 and were receiving two divided daily doses of tacrolimus in their initial regimen for prevention of allograft rejection
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Trough tacrolimus blood concentration to dose ratio | 3 days after transplant

SECONDARY OUTCOMES:
Proportion achieved the target trough blood concentration within the first week | 7 days after transplant
Acute rejection rate | 3 months after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Chagriya Kitiyakara, MD, Study Chair — Ramathibodi Hospital, Faculty of Medicine, Mahidol University

REFERENCES:
- [Derived] Yaowakulpatana K, Vadcharavivad S, Ingsathit A, Areepium N, Kantachuvesiri S, Phakdeekitcharoen B, Sukasem C, Sra-Ium S, Sumethkul V, Kitiyakara C. Impact of CYP3A5 polymorphism on trough concentrations and outcomes of tacrolimus minimization during the early period after kidney transplantation. Eur J Clin Pharmacol. 2016 Mar;72(3):277-83. doi: 10.1007/s00228-015-1990-0. Epub 2015 Dec 4. PMID 26635230